CLINICAL TRIAL: NCT05697614
Title: The Efficacy and Safety of First-Line Anti-Epileptic Drugs (AEDs) as Substitution Therapy in Children Who Are Resistant to Second-Line AEDs
Brief Title: The Benefit and Safety of Older Generation Anti-Epileptic Drugs (AEDs) in Drug-Resistant Epilepsy Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Roro Rukmi Windi Perdani, Principal investigator, Dr Cipto Mangunkusumo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-09-1097
Record Dates: First submitted 2022-11-28; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Drug Resistant Epilepsy
Keywords: anti-epilepsy drug; children; epilepsy; resistant
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsy | interventions — Valproic Acid; Carbamazepine; Phenytoin; Lamotrigine; Clobazam; Oxcarbazepine

STUDY DESIGN:
Intervention Model Description: The subjects will be randomized into 2 groups : intervention and control. The subjects will be recruited by consecutive sampling technique
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): valproic acid 15 - 60 mg/kg body weight/day, divided into 2 dosages/day for 12 weeks ; carbamazepine 10 - 30 mg/kg body weight/day, divided into 2 dosages/day for 12 weeks ; phenytoin 5-7 mg/kg body weight/day, divided into 2 dosages/day for 12 weeks
  Interventions: Drug: Valproic acid; Drug: Carbamazepin; Drug: Phenytoin
- control (Active Comparator): lamotrigine 0.2 mg/kg body weight/day, divided into 2 dosages/day for 12 weeks ; clobazam 0.1 - 0.8 body weight/day, divided into 2 dosages/day for 12 weeks ; oxcarbazepine10 - 30 mg/kg body weight/day, divided into 2 dosages/day for 12 weeks
  Interventions: Drug: Lamotrigine; Drug: Clobazam; Drug: Oxcarbazepine

INTERVENTIONS:
Drug: Valproic acid — valproic acid is used for general epilepsy type, used in experimental group
  Other Names: sodium divalproex; depaken
  Arms: intervention
Drug: Carbamazepin — carbamazepine is used for focal type epilepsy, used in experimental group
  Other Names: tegretol; bamgetol
  Arms: intervention
Drug: Phenytoin — phenytoin is used for both general or focal epilepsy in case valproic acid or carbamazepine is contraindicated, used in experimental group
  Other Names: kutoine
  Arms: intervention
Drug: Lamotrigine — lamotrigine is used for general epilepsy type, used in control group
  Other Names: lamictal
  Arms: control
Drug: Clobazam — clobazam is used for both general or focal epilepsy in case if lamotrigine or oxcarbazepine is not possible to be administered and is used particularly in myoclonic jerk , used in control group
  Other Names: frisium
  Arms: control
Drug: Oxcarbazepine — oxcarbazepine is used for focal type epilepsy, used in control group
  Other Names: trileptal
  Arms: control

SUMMARY:
The goal of this interventional study is to learn about the efficacy and safety of first line anti epileptic drugs (AEDs) as substitution therapy for children who are resistant to second-line AEDs. The main question to answer it aims are :

how much the difference proportion of responders (responders are children who achieve the decrease of seizure frequencies by 50%) how much time it is needed to achieve the decrease of seizure frequencies by 50% The patients who are eligible for the study and have given their consent, will be enrolled, divided into 2 groups, the control and intervention.

The participant should follow the 14 weeks of intervention that consists of 6 phases : baseline, initial dose, titration dose, maintenance dose, tapering-off dose, and new combination maintenance dose.

DETAILED DESCRIPTION:
Each phase of the study is described below

In baseline phase, data such as demographic, clinical characteristic including seizure frequency, seizure type, seizure onset, medication history, family history of seizure, and also developmental stages, will be recorded from electronic medical record. Besides, the CT-scan or MRI are also collected from the same source. After that, their quality of life will be assessed by QOLCE-55 validated questionnaire through self-guided report. Furthermore, the laboratory investigation and EEG will be performed.

The next phase is intervention phase, started from initial phase and ended by the maintenance of new combination therapy phase, takes with overall 12 weeks. Initially, the substitution drugs with each initial dose are consumed. The drugs consist of valproic acid for the generalized and carbamazepine for focal epilepsies.

On the other hand, the control group will take lamotrigine or clobazam for generalized and oxcarbazepine for focal ones. The phase continuous to titration dose, in which, the dose is raised gradually until it causes 50% of seizure reduction, and the next step is maintained the dose for about 2 weeks.

- The following is tapering-off and after that stopping the substituted drug, levetiracetam or topiramate, which is determined by considering individual condition. Yet, if the seizures increase more than one and a half time of the previous frequency during the phases, the intervention will be ended immediately. On the contrary, if the condition is better, then the children go to the maintenance of new combination, that is the substitution drug and the old drugs in which the seizures do not go up or even better keep going down.

ELIGIBILITY:
Inclusion Criteria:

1. Children age at 1 - 18 years old
2. Children diagnosed as drug-resistant epilepsy by pediatric neurologists, diagnosis was based on the ILAE 2017 criteria
3. Children will have got at least 3 months of combination therapy that consists of levetiracetam of topiramate with optimal dosage but haven't got seizure reduction

Exclusion Criteria:

1. Non-convulsive epilepsy
2. Suffered from status epilepticus in the prior 3 months before the study begins Past medical history of idiosyncrasies or severe adverse drug reactions caused by the
3. substitution therapy that will be given

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
the different proportion of responders between groups who get first-line anti-epileptic drugs (intervention) and second-line anti-epileptic drugs (control) | trough the study completion, about 14 weeks
  responders are children who get the reduction of seizure frequency by 50%

SECONDARY OUTCOMES:
time to achieve the reduction of seizure frequency by 50% or more among responders | during intervention, about 12 weeks
  time that is counted in week and is divided into 3 categories , 2-<4 weeks, 4-<8 weeks and 8-12 weeks
the difference of quality of life between groups who get first-line anti-epileptic drugs (intervention) and second-line anti-epileptic drugs (control) | at baseline phase in the 1st week (before intervention) and after intervention in the 14th week
  quality of life is assessed by validated instrument QOLCE-55. It has 55 questions including cognitive (22 items), emotional (17 items), social (7 items) and also physical (9 items) function. Items are rated on a five-point Likert scale, 0 = very often, 1 = fairly often, 2 = sometime, 3 = almost never, 5 = never. The composite score is the unweighted average of the four subscales, ranging from 1-100, higher score indicates better quality of life. b. Differences in quality of life: quality of life assessment using QOLCE-55 instrument. The average of each function (cognitive, emotional, social and physical functions) and the average of the total functions are assessed. This variable is categorized into:
  * Different, if there is a difference in the average quality of life
  * Not different, if there is no difference in the average quality of life
the difference of the electroencephalography (EEG) changing between groups who get first-line anti-epileptic drugs (intervention) and second-line anti-epileptic drugs (control) | at baseline phase in the 1st week (before intervention) and after intervention in the 14th week
  The EEG examination is operated two times, at the baseline and post intervention phase, with high density machine (Caldwell Easy III) is done twice, pre- and post-intervention. The machine will operate for about 45 minutes including 5 minutes each for eye-open and eye-close in every subjects. Beginning with acquisition, EEG recordings use standard parameter to analyze brain activity at various frequencies to gain good quality and artefact-free result. The printed results of the EEG is available for about 4-7 days after the examination.
  EEG recording results are categorized into:
  * Normal : does not show of hypofunction/asymmetry/epileptiform waves
  * Abnormal: shows a picture of hypofunction/asymmetry/epileptiform waves or a combination of 1 or more of these features The subjects who show changes in their EEG are later grouped into groups of abnormal to normal or abnormalities that showed improvement. Abnormalities that show improvement, for example are hypofunction (slowing down)
the description of age in percentage | at baseline phase in the 1st week (before intervention)
  the data is taken from electronic medical record, age is categorized into <5 years, 5-<10 years, and >/= 10 years
the description of seizure onset in percentage | at baseline phase in the 1st week (before intervention)
  the data is taken from electronic medical record, seizure onset is categorized into <5 years, 5-<10 years, and >/= 10 years
the description of gender in percentage | at baseline phase at 1st week (before intervention)
  the data is taken from electronic medical record, gender is categorized into male and female
the description duration of anti epileptic drug medication | at baseline phase at 1st week (before intervention)
  the data is taken from electronic medical record, the duration is categorized into <1 year , 1 - <2 year, 2 - 5 year, and > 5 year
The brain CT or brain MRI | at baseline phase at 1st week (before intervention)
  The brain CT or brain MRI are taken from electronic medical record, categorized into normal and abnormal findings. it is categorized as normal if the brain, liquor cerebrospinal and skull is within normal range (no deformation of skull, no hydrocephalus, the brain volume is normal, and no signs of infection such as enhancement, no hemorrhage, no calcification)
The adverse drug reaction profile in percentage | during intervention, about 12 weeks
  The adverse drug reaction profile are taken from the diary card, it is categorized into neurology system, gastrointestinal system, musculocutaneous system, renal function, liver function and electrolyte
seizure frequency | during intervention, about 12 weeks
  the frequency is how many times in a month, it is categorized into <5 times, 5-10 times, 10-20 times and > 20 times
the history of developmental delayed | at baseline phase at 1st week (before intervention)
  the data is taken from electronic medical record, categorized into yes or no. it is named as delayed if the development does not follow the milestone in one or more developmental sectors (language, gross motor skill, fine motor skill, personal social)
the number of anti-epileptic drug is consumed | at baseline phase at 1st week (before intervention)
  the data is taken from electronic medical record, it is categorized into 2 , 3 , or >3 drugs
the history of seizure in the family | at baseline phase at 1st week (before intervention)
  the data is taken from electronic medical record, it is categorized into yes or no
the association between age and seizure reduction | after intervention in the 14th week
  the age is categorized into <5 years, 5-<10 years, and >/= 10 years ; seizure reduction is categorized into responder and non-responder
the association between seizure onset and seizure reduction | after intervention in the 14th week
  seizure onset is categorized into <5 years, 5-<10 years, and >/= 10 years ; seizure reduction is categorized into responder and non-responder
the association between gender and seizure reduction | after intervention in the 14th week
  gender is categorized into male and female ; seizure reduction is categorized into responder and non-responder
the association between duration of anti epileptic drug medication and seizure reduction | after intervention in the 14th week
  he duration is categorized into <1 year , 1 - <2 year, 2 - 5 year, and > 5 year ; seizure reduction is categorized into responder and non-responder
the association of the brain CT or brain MRI and seizure reduction | after intervention in the 14th week
  the brain CT or brain MRI categorized into normal and abnormal findings. it is categorized as normal if the brain, liquor cerebrospinal and skull is within normal range (no deformation of skull, no hydrocephalus, the brain volume is normal, and no signs of infection such as enhancement, no hemorrhage, no calcification). Seizure reduction is categorized into responder and non-responder
the association of seizure frequency and seizure reduction | after intervention in the 14th week
  the frequency is how many times in a month, it is categorized into <5 times, 5-10 times, 10-20 times and > 20 times. Seizure reduction is categorized into responder and non-responder
the association between the history of developmental delayed and seizure reduction | after intervention in the 14th week
  the history of developmental delayed is categorized into yes or no. it is named as delayed if the development does not follow the milestone in one or more developmental sectors (language, gross motor skill, fine motor skill, personal social). Seizure reduction is categorized into responder and non-responder
the association of the number of anti-epileptic drug is consumed and seizure reduction | after intervention in the 14th week
  number of anti-epileptic drug consumed is categorized into 2 , 3 , or >3 drugs. Seizure reduction is categorized into responder and non-responder
the association between the history of seizure in the family and seizure reduction | after intervention in the 14th week
  the history of seizure in the family is categorized into yes or no. Seizure reduction is categorized into responder and non-responder

CONTACTS AND LOCATIONS:
Overall Officials: Roro Rukmi Windi Perdani Pediatrician, Principal Investigator — Cipto Mangunkusumo Hopsital - Medical Faculty of Indonesia University
Locations (3):
- Indonesia (3):
  - Cipto Mangunkusumo Hospital, Jakarta Pusat, Jakarta Special Capital Region
  - Harapan Kita Hospital, Jakarta
  - Fatmawati Hospital, Jakarta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perdani RRW, Arozal W, Mangunatmadja I, Kaswandani N, Handryastuti S, Medise BE, Hardi H, Thandavarayan RA, Oswari H. The efficacy and safety of first-line anti-seizure medications as substitution therapy for children with drug-resistant epilepsy: a randomized controlled trial protocol. Front Neurol. 2023 Aug 7;14:1237183. doi: 10.3389/fneur.2023.1237183. eCollection 2023. PMID 37609651

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-09-29): https://cdn.clinicaltrials.gov/large-docs/14/NCT05697614/Prot_SAP_ICF_000.pdf